CLINICAL TRIAL: NCT06527001
Title: Retrospective Analysis of Mesenteric Lymph Node Metastasis and Nutritional Status After Bowel Resection for Ovarian Cancer
Brief Title: Mesenteric Lymph Node Metastasis and Nutritional Status After Bowel Resection for Ovarian Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Ying Zhou-1
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Progression-Free Survival; Overall Survival; Nutrition Aspect of Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Residual Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is an observational study and did not involve interventions.

SUMMARY:
Ovarian cancer is one of the three major malignant tumors in gynecology, causing more than 200,000 deaths globally each year, with the highest mortality rate. However, due to its insidious onset and lack of specificity in clinical manifestations, nearly 70% of patients are in advanced stages upon diagnosis. Ovarian cancer often spreads along the peritoneal surface of the abdominal and pelvic cavity and involves the intestines through direct extension or plasma membrane infiltration, resulting in impaired intestinal function and intestinal obstruction. Cytoreductive Surgery is a critical treatment for patients with ovarian cancer. Literature reports that about 60%-70% of patients with advanced ovarian cancer underwent bowel resection at the time of primary debulking surgery, with the main site of resection being the recto-sigmoid (48%-55%), followed by the rest of the colon (18%-20%) and the small bowel (6%-27%). Patients with bowel resection for ovarian cancer often have involvement of mesenteric lymph nodes (MLN), and the positive rate of MLN fluctuates from 37% - 79.4%, and the incidence of liver metastasis within 3 years in ovarian cancer patients with MLN involvement is 61.1%. However, ovarian cancer patients with bowel or liver involvement are susceptible to postoperative malnutrition due to their extensive surgery, as well as increased incidence of postoperative complications. Therefore, this study included patients who underwent bowel resection for ovarian cancer, and assessed the patients' MLN metastasis and nutritional status based on the relevant clinical indicators, in order to reduce the incidence of postoperative complications in patients with bowel resection, to improve the patients' prognosis, and to enhance the quality of life.

DETAILED DESCRIPTION:
This is a non-interventional retrospective study to collect clinical data from patients with advanced epithelial ovarian cancer who underwent bowel surgery in the Department of Obstetrics and Gynecology of the First Affiliated Hospital of the University of Science and Technology of China from January 2017 to December 2023. The information collected includes: age, preoperative body mass index (BMI), menopausal status, genetic test results, FIGO stage, type of bowel resection, duration of the operation, and depth of bowel infiltration, number of MLN resections, as well as nutritional status scores (NRS 2002 and PG-SGA), biochemical indices (serum albumin, prealbumin, total protein and so on), inflammatory indices (C-reactive protein, neutrophilic to lymphocyte ratio, platelet to lymphocyte ratio), and anthropometric parameters (body weight change, BMI). The aim of the clinical data analysis was to reduce the incidence of perioperative complications, improve the prognosis, and enhance the quality of life of patients with ovarian cancer after bowel surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced epithelial ovarian cancer who underwent bowel surgery (PDS, IDS, and SCS);

  * FIGO (2014) staging of stage III to IV;

    * Diagnosis was made between January 2017 and December 2023; ④Complete relevant clinical data.

Exclusion Criteria:

* Combination of malignant tumors in other parts of the body not in remission or under treatment; ②Having an infectious disease in the infectious or active stage;

  * Unknown status of visits to other hospitals and loss of visits; ④Not considered by the investigator to be suitable for enrollment or incomplete baseline information.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a non-interventional retrospective study to collect clinical data from patients with advanced epithelial ovarian cancer who underwent bowel surgery in the Department of Obstetrics and Gynecology of the First Affiliated Hospital of the University of Science and Technology of China from January 2017 to December 2023.All enrolled patients underwent cytoreductive surgery and completed follow-up registration according to NCCN guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 year
  PFS is defined as the time interval between a patient's diagnosis of gynecological malignancy and the first occurrence of progression of the disease or death from any cause.
OS | 2 year
  OS was defined as the time interval between a patient's diagnosis of gynecologic malignancy and death from any cause or the end of the last follow-up date.
NRS 2002 | The scale was evaluated before surgery and at 4 months after surgery.
  Nutritional Risk Screening 2002 (NRS 20002) was primarily used to assess a patient's possible nutritional risk, and a score of ≥3 indicates that the patient is at risk of malnutrition or nutritional risk.
PG-SGA | The scale was evaluated before surgery and at 4 months after surgery.
  Patient-Generated Subjective Global Assessment (PG-SGA) was primarily used to assess the nutritional status of tumor patients. Well nourished was 0-1 score, suspected or mild malnutrition was 2-3 score, moderate malnutrition was 4-8 score, severe malnutrition ≥9 score.
BMI | The index was evaluated before surgery and at 4 months after surgery.
  Body mass index (BMI) was obtained by dividing weight in kilograms by height in meters squared. Normal was 18.5-24 score, overweight was 24-28 score, and obesity ≥28 score.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhou, MD, Study Chair — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Locations (1):
- Anhui Provincal Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No